CLINICAL TRIAL: NCT03068247
Title: Neurobiology of Non-Specific and Specific Treatment Responses in Major Depression
Brief Title: Neurobiology of Treatment Responses in MDD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Institution was unable to manufacture radiotracer that was central to the protocol. Study transferred to another institution.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 00095062
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): 10 weeks of duloxetine beginning at 30 mg per day for week 1, then 60 mg / day thereafter.
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): 10 weeks of placebo once daily for 1 week, then twice daily therafter.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 10 week treatment
  Other Names: Cymbalta
  Arms: Interventional
Drug: Placebo — 10 week treatment
  Arms: Placebo

SUMMARY:
The primary study intent is to examine biological mechanisms associated with acute and chronic treatment responses in major depressive disorder (MDD). It is hypothesized that treatment responsiveness, representing endogenous opioid system function, will be associated with acute improvements in mood state over a 10-week treatment trial in MDD. Potential (bio) markers of treatment effects will be tested against psychophysical responses to placebo and active treatments.

DETAILED DESCRIPTION:
Volunteers will be randomized to receive placebo pills or a commercially available SNRI for 10 weeks. Volunteers will undergo imaging with structural and functional MRI and PET with [11C]carfentanil to determine baseline μOR BPND and changes in BPND measures during acute i.v. medication administration at the time of scanning before and after the 10-week treatment period.

To elicit the activation of µ-opioid-mediated neurotransmission in the scanner, we utilize the introduction of medication (active or inactive) 1mL into an intravenous port every 4 minutes, 15 sec per infusion, starting 45 minutes after radiotracer administration, until scan completion. Participants are made aware that the study drug will be administered at the time a computer-generated human voice recording reads a second-by-second count of the infusion timing (15 sec).

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM V criteria for Major Depressive Episode, single episode or recurrent, for at least a month;
* Unmedicated for at least 10 half-lives of the previous AD used;
* Willing to limit the introduction of any new treatments during the study;
* 18 - 55 years of age;
* Right handed;
* Capable of giving written informed consent;
* Hamilton Depression Rating Scale (17-item HDRS, not including atypical features) >15 at screening and randomization;

Exclusion Criteria:

* Major medical illness (e.g., cancer, HIV, Hepatitis C, etc.) or concurrent, untreated, or symptomatic medical illnesses, including acute or ongoing pain, autoimmune or inflammatory disease;
* Use of narcotic analgesics within the last 6 months or regular use of sleeping aids (including benzodiazepines and related compounds), more than twice a week;
* Recent history of substance abuse (within the last 6 months) or history of substance dependence (lifetime);
* Other comorbid psychiatric illnesses, such as Bipolar Disorder, Obsessive Compulsive Disorder, Panic Disorder, any psychosis, or Axis II diagnoses. Generalized Anxiety and Social Anxiety Disorders will NOT be considered exclusionary given their common association with MDD
* Concurrent participation in other therapeutic trials;
* Pregnancy/nursing;
* Ongoing treatment with medications with psychotropic properties;
* Contraindications to PET or MRI methods;
* Impairments, activities or situations that would prevent completion of the study protocol;
* Prior non-response to duloxetine;
* Active suicidal ideation.
* Urine screens positive for opioids or any substances of abuse.
* Allergy to fentanyl (because of structural similarity to the radiotracer [11C]carfentanil to be employed in the study).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
mu-opioid receptor binding capacity | 10 weeks
  derived from PET scans
depression score | 10 weeks
  HRSD-17 score

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No